CLINICAL TRIAL: NCT00084773
Title: A Pilot Clinical Trial of Preoperative Cetuximab With Concurrent Continuous Infusion Fluorouracil and Pelvic Radiation in Patients With Local-Regionally Advanced Rectal Cancer
Brief Title: Neoadjuvant Cetuximab, Fluorouracil, and Pelvic Irradiation in Treating Patients With Locally Advanced or Locally Recurrent Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-006; MSKCC-04006
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Cancer
Keywords: recurrent rectal cancer; stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Fluorouracil; Neoadjuvant Therapy; Radiotherapy

ARMS (1):
- Cetuximab, Fluorouracil, and Pelvic Irradiation (Experimental): Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, 43, 50, 57, and 64 and fluorouracil IV continuously on days 1-42. Patients undergo whole-pelvic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Approximately 1-3 weeks after completion of study treatment, patients undergo surgical resection followed by adjuvant chemotherapy off-study.
  Patients are followed for up to 5 years.
  Interventions: Biological: cetuximab; Drug: fluorouracil; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab
Drug: fluorouracil
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies such as cetuximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy such as fluorouracil work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving cetuximab with fluorouracil and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety profile of neoadjuvant cetuximab, fluorouracil, and pelvic irradiation in patients with locally advanced or locally recurrent rectal cancer.

Secondary

* Determine the activity of this regimen, in terms of pathological complete response rate, in these patients.

OUTLINE: This is a non-randomized, open-label, pilot study.

Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, 22, 29, 36, 43, 50, 57, and 64 and fluorouracil IV continuously on days 1-42. Patients undergo whole-pelvic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-40. Treatment continues in the absence of disease progression or unacceptable toxicity.

Approximately 1-3 weeks after completion of study treatment, patients undergo surgical resection followed by adjuvant chemotherapy off-study.

Patients are followed for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed rectal adenocarcinoma meeting 1 of the following staging criteria:

  * Locally advanced disease

    * Resectable (uT3) disease

      * Primary gross transmural tumor that is not adherent to adjacent pelvic structures by endorectal ultrasound
    * Primary tethered or unresectable (cT4 or uT4) disease

      * Primary tumor is contiguous with or adherent or fixed to adjacent pelvic structures by clinical exam and CT scan
      * Primary surgery would likely leave residual tumor
    * Small volume extrapelvic metastases allowed
  * Recurrent disease after definitive resection

    * Disease limited to the pelvis
* Requires combined modality treatment
* Epidermal growth factor receptor status-positive, -negative, or -unknown
* If previously treated with adjuvant fluorouracil-based chemotherapy, no disease recurrence during or within 12 months after completion of adjuvant therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0 -1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin > 8.0 g/dL
* Platelet count > 150,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine ≤ 1.5 times upper limit of normal

Cardiovascular

* No myocardial infarction within the past 6 months
* No evidence of uncontrolled congestive heart failure requiring therapy

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No known severe hypersensitivity to cetuximab or any of its excipients
* No uncontrolled infection
* No high-grade bowel obstruction (bowel lumen ≤ 1 cm) unless patient has undergone protective surgical diversion or endoscopic stenting procedure
* No other concurrent medical or psychiatric condition or disease that would preclude study participation
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior cetuximab
* No prior murine or chimeric monoclonal antibody therapy
* No prior biological response modifiers for metastatic colorectal cancer
* No concurrent anti-vascular endothelial growth factor/Flk-1 monoclonal antibody therapy
* No other concurrent antibody therapy or immunotherapy
* No concurrent gene therapy
* No concurrent vaccine therapy
* No concurrent angiogenesis inhibitors, including thalidomide

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy for metastatic colorectal cancer
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* No prior radiotherapy for metastatic colorectal cancer
* No prior pelvic radiotherapy
* No other concurrent radiotherapy

Surgery

* See Disease Characteristics
* Fully recovered from prior oncologic or other major surgery

Other

* No other prior therapy that targets the epidermal growth factor receptor pathway
* No other concurrent experimental therapy or drugs
* No concurrent matrix metalloprotease inhibitors
* No concurrent participation in another clinical study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-03; Primary Completion 2007-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety profile | 2 years

SECONDARY OUTCOMES:
Activity in terms of pathological complete response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States